CLINICAL TRIAL: NCT06163053
Title: A French Non-interventional Prospective Multicenter Study Evaluating Quality of Care Perception of Cancer Patients Treated by Immunotherapy at Home - SATISFACT-HOME
Brief Title: A Study to Evaluate Satisfaction With Care in Patients With Cancer Receiving Immunotherapy Treatment at Home
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-6JE
Record Dates: First submitted 2023-11-30; First posted 2023-12-08 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Cancer; Solid Tumors
MeSH Terms: conditions — Neoplasms | interventions — Immunotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants receiving immunotherapy at home
  Interventions: Drug: Immunotherapy

INTERVENTIONS:
Drug: Immunotherapy — Immune checkpoint inhibitors in approved indications

SUMMARY:
The purpose of this observational study in France is to evaluate changes in satisfaction with care in participants with solid tumors who transitioned from receiving immunotherapy treatment in the hospital outpatient setting to receiving treatment at home

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years old
* Participants whose oncology specialist has already initiated treatment with immune checkpoint inhibitors (ICIs) in the outpatient hospital setting for an advanced solid tumor (as monotherapy or in combination) or as adjuvant therapy, in an indication approved and reimbursed in France
* Participants whose oncology specialist has independently of the study defined their eligibility for hospital at home (HAH) before contacting the HAH unit for final admission
* Participants who provide oral informed consent to participate in the study

Exclusion Criteria:

* Participants who have expressed an opposition to their data collection
* Participants under guardianship
* Participants taking part in an interventional study for cancer treatment with at least one ICI as an investigational drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants in France with solid tumors transitioning from receiving immunotherapy treatment in the hospital outpatient setting to receiving treatment at home
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2023-08-29 (Actual); Primary Completion 2025-06-12 (Actual); Study Completion 2025-06-12 (Actual)

PRIMARY OUTCOMES:
Change in patient satisfaction on the European Organisation for Research and Treatment of Cancer satisfaction with cancer care core questionnaire (EORTC PATSAT-C33) when transitioning from Outpatient Hospital to Hospital at Home to receive immunotherapy | Participants follow up approximately 24 weeks after transition to treatment at home

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (3):
- France (3):
  - CH Metropole Savoie, Chambéry
  - CH Francois Quesnay, Mantes-la-Jolie
  - CH de Pau, Pau

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm